CLINICAL TRIAL: NCT04548765
Title: Evaluation of Letters Enhanced With Behavioral Nudges to Promote Colorectal Cancer Testing Through Fecal Immunochemical Tests or Colonoscopies
Brief Title: Evaluation of Letters Promoting Colorectal Cancer Testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Responsible Party: Principal Investigator, Amir Goren, Program Director, Behavioral Insights Team, Geisinger Clinic
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Screening
Other Study IDs: 2020-0510
Record Dates: First submitted 2020-09-04; First posted 2020-09-16 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-09

CONDITIONS: Cancer Colorectal
Keywords: Mass Screening; Communication; Occult Blood; Colonoscopy; Risk Reduction Behavior; Economics, Behavioral; Psychology; Loss Framing; Fear Appeals; Default Effect; Decoy Effect
MeSH Terms: conditions — Colonic Neoplasms; Communication; Risk Reduction Behavior; Behavior | interventions — College Fraternities and Sororities; Price Transparency

STUDY DESIGN:
Intervention Model Description: 1 x 4 design
Who Masked: Participant, Care Provider
Masking Description: Participants and providers are not aware of the different letter versions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard Letter (Active Comparator): The standard letter describes the importance of getting screened and instructs recipients how to use the FIT kit for screening at home.
  Interventions: Behavioral: Letter
- Letter with Risks (Experimental): The standard letter is enhanced with language that further emphasizes the risks but also clearly describes how early detection with a test can reduce those risks; it also explains why test kits are being sent to disarm skepticism about the program.
  Interventions: Behavioral: Letter; Behavioral: Loss Frame and Fear Appeals; Behavioral: Transparency
- Letter with Risks and Options (Experimental): In addition to the enhancements added by the letter with risks, the letter also includes a table comparing FIT kit and colonoscopy. Presenting different screening options allows recipients to make the choice that best suits them. In addition, presenting multiple options increases the chance that recipients get screened in one way or another.
  Interventions: Behavioral: Letter; Behavioral: Loss Frame and Fear Appeals; Behavioral: Default Effect and Presentation of Alternatives; Behavioral: Enhanced Fear Appeals and Decoy Effect
- Letter with Risks, Options, and Consequences for Inaction (Experimental): In addition to the enhancements added by the letter with risk, the comparison table includes comparisons of the consequences of getting screened vs. waiting for symptoms to appear.
  Interventions: Behavioral: Letter; Behavioral: Loss Frame and Fear Appeals; Behavioral: Enhanced Fear Appeals and Decoy Effect

INTERVENTIONS:
Behavioral: Letter — Recipients receive a letter promoting CRC screening.
Behavioral: Loss Frame and Fear Appeals — The letter is enhanced with language that frames the situation in terms of losses. It also uses fear appeals by showing the risks of colorectal cancer, while also showing that screening is an achievable means to address those risks.
  Arms: Letter with Risks; Letter with Risks and Options; Letter with Risks, Options, and Consequences for Inaction
Behavioral: Transparency — The letter explains why the kit was sent, which makes the purposes of the mailing clear to the recipient.
  Arms: Letter with Risks
Behavioral: Default Effect and Presentation of Alternatives — The pros and cons for screening with FIT kits and colonoscopy are presented. By showing an additional option, the table frames the FIT kit as the default option (since they are included in the mailer). In this situation, inaction is no longer the default option. Changing the default option increases the chance that the FIT kit is used. In addition, another viable alternative is provided (colonoscopy), which still contributes to the goal of the project (getting screened).
  Arms: Letter with Risks and Options
Behavioral: Enhanced Fear Appeals and Decoy Effect — Comparisons of the mortality rates between screening with FIT kits, colonoscopy, and inaction (waiting for symptoms to appear) are displayed. Inaction is presented as a decoy, which has worse outcomes than either of the screening options. Due to this contrast, the inclusion of the decoy increases the appeal of the other screening options.
  Arms: Letter with Risks and Options; Letter with Risks, Options, and Consequences for Inaction

SUMMARY:
In this evaluation, 4 different versions of letters are being sent with mailers promoting colorectal cancer screening with an at-home test. The researchers hypothesize that the use of behavioral nudges in the message should lead to increased colorectal cancer screening (either with the at-home test or a colonoscopy).

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the third most common cancer diagnosed in the US. Mailing fecal immunochemical (FIT) kits to at-risk patients is an effective way of increasing CRC testing uptake, as this test can be done at home and is less intrusive compared to colonoscopies. As part of an existing program, the health system mails FIT kits to eligible patients each year. Although this test needs to be conducted annually, not everyone who receives the test kit returns the kits for processing. In this study, the researchers aim to test different letters with the goal of encouraging the use of FIT kits or scheduling a colonoscopy.

As part of this study, the kits are mailed with everything the patient will need to conduct the test at home and mail a sample back to the hospital. It also includes an introductory letter informing the patient about the program and inviting them to use the kit. The researchers are comparing a standard version of the introductory letter against 3 versions that include different combinations of behavioral nudges, specifically framing effects (loss, default, decoy) and fear appeals.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment in Medicare Health Maintenance Organization (HMO) and Preferred Provider Organization (PPO; age 65 and older) or Commercial HMO in one large employer's group
* Has a flag indicating that the person is due for a colon cancer screening

Exclusion Criteria:

- Members who are on the do not contact list at Geisinger Health Plan

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14644 (Actual)
Dates: Start 2020-07-24 (Actual); Primary Completion 2021-01-24 (Actual); Study Completion 2021-07-23 (Actual)

PRIMARY OUTCOMES:
FIT Kit Return at 6 months | 6 months from intervention start date
  Binary variable indicating whether a valid FIT kit was returned for testing
Colonoscopy Ordered at 6 months | 6 months from intervention start date
  Binary variable indicating whether a colonoscopy was ordered

SECONDARY OUTCOMES:
FIT Kit Return at 12 months | 12 months from intervention start date
  Binary variable indicating whether a valid FIT kit was returned for testing (a longer time frame allows for late responses)
Colonoscopy Ordered at 12 months | 12 months from intervention start date
  Binary variable indicating whether a colonoscopy was ordered (a longer time frame allows for late responses)
FIT Kit Result | 12 months from intervention start date
  Binary variable indicating whether the test was positive or negative (if FIT kit was returned)
Colonoscopy Completed | 12 months from intervention start date
  Binary variable indicating whether the colonoscopy was completed (if colonoscopy was ordered)
Colonoscopy Result | 12 months from intervention start date
  Binary variable indicating whether the test was positive or negative (if colonoscopy was completed)

CONTACTS AND LOCATIONS:
Overall Officials: Amir Goren, PhD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data with no personally identifiable information will be made available to other researchers on the Open Science Framework for transparency. This will include the essential data and code needed to replicate the analysis that yielded reported findings. The PI did not examine or analyze any data from this study prior to this registration.
Supporting Information: Study Protocol, Analytic Code
Time Frame: The data will become available after publication of study results in a scientific journal and will be available as long as the Open Science Framework hosts the data.
Access Criteria: The data on the Open Science Framework will be open to anyone requesting that information.
URL: http://osf.io

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-16): https://cdn.clinicaltrials.gov/large-docs/65/NCT04548765/Prot_SAP_000.pdf